CLINICAL TRIAL: NCT07009327
Title: Efficacy and Safety of Photodynamic Therapy for Cervical Intraepithelial Neoplasia 3(CIN3):A Multicenter Prospective Cohort Study
Brief Title: Efficacy and Safety of Photodynamic Therapy for CIN3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDT-CIN3; 2022YFB3604704 (Other Grant/Funding Number: Ministry of Science and Technology of the People's Republic of China)
Record Dates: First submitted 2025-05-13; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Precancerous Cervical Lesion
Keywords: PDT; HPV; CIN 3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALA-PDT (Other): Patients choose PDT to treat the disease
  Interventions: Procedure: ALA-PDT

INTERVENTIONS:
Procedure: ALA-PDT — use ALA_PDT to treat the disease

SUMMARY:
To investigate the efficacy and safety of photodynamic therapy (20% 5-amino-ketovalerate 630nm red light) in the treatment of cervical intraepithelial neoplasia 3(CIN 3)in women in the real world

ELIGIBILITY:
Inclusion Criteria:

* CIN3, photodynamic therapy was required,
* type 1 2 transformation area, colposcopy was sufficient
* the lesion boundary was completely visible
* The ECC did not indicate high-grade lesions

Exclusion Criteria:

* coexistence or suspicion of cancer;
* TCT HSIL
* involving glands
* Porphyria patients, or suspected allergic to red and blue light.
* severe medical comorbidities；

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the treatment | 1 month after the treatment
  colposcopy and biopsy will be performed one month after the treatment. Patients will be categorised as having complete remission(CR) if biopsy confirmed LSIL. If CIN 2 was found after the first course of PDT, it would be categorised as partial remission(PR). Those with the same grade were categorised as persistent disease(PD).
  The proportion of CR after PDT treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Qin Han, Study Chair — Peking Unniversity Third Hospital
Locations (1):
- Peking Unniversity Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Chinese women attach great importance to privacy issues related to sex and do not accept the disclosure of their information

DOCUMENTS (2):
  • Study Protocol (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT07009327/Prot_000.pdf
  • Informed Consent Form (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT07009327/ICF_001.pdf